CLINICAL TRIAL: NCT00918372
Title: Coronary Atherosclerosis in Women Athletes: Asymptomatic Twin Cities Marathon Women Studied by MSCT Angiography
Brief Title: Coronary Artery Disease (CAD) in Women Marathon Runners
Status: Completed | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Robert Stockton Schwartz, Minneapolis Heart Institute Foundation
Other Study IDs: img001
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Coronary Artery Disease
Keywords: MSCTA; Marathon runners
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Extreme fitness: Female competitive long distance runners
- Control: Age and Risk matched controls

SUMMARY:
The aim of this study is to determine the effects of extreme fitness in women. The incidence of coronary artery disease observed via multislice computed tomography (MSCT) angiogram will be compared with age and risk-matched controls from both sedentary and fitness activity groups who have never been significant runners. Life style, training volume and risk factors will be assessed.

DETAILED DESCRIPTION:
Single-center, non-randomized, prospective, observational study. The study population will be up to 100 female athletes who are competitive long distance runners, and have been so for a minimum of 10 years. Multi-slice computed tomography (MSCT) will be used to characterize the amount, severity and type of atherosclerotic lesions. MSCTA will be performed per usual practice using a minimum X-ray dose protocol.

The study will determine whether moderate to high intensity, long term athletic training and competition is associated with enhanced coronary artery disease in women. Each participant will complete a life-style, training volume and risk factor questionnaire. These participants will be compared to an age, gender and risk factor matched cohort.

ELIGIBILITY:
Inclusion Criteria:

* Female athletes who have run marathons competitively for a minimum of 10 years.
* Age > 40 years old
* Agree to participate and sign an informed consent form

Exclusion Criteria:

* Allergy to X-ray contrast
* Creatinine ≥ 2.0
* Pregnant Female
* Has run a marathon within the past 2 weeks

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female long distance runners as compared to age and risk-matched controls from both sedentary and fitness activity groups who have never been significant runners, derived from the Minneapolis Heart Institute Foundation's (MHIF) Cross-Sectional Imaging database.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Evidence of coronary artery disease confirmed by Multislice Computed Tomography | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Schwartz, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Minneapolis Heart Institute at Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Angeli SJ, Haft JI. Severe coronary artery disease in a marathon runner. Chest. 1987 Feb;91(2):271-2. doi: 10.1378/chest.91.2.271. PMID 3802941
- [Background] Bassler TJ. Coronary-artery disease in marathon runners. N Engl J Med. 1980 Jan 3;302(1):57-8. No abstract available. PMID 7350403
- [Background] Colt E. Coronary-artery disease in marathon runners. N Engl J Med. 1980 Jan 3;302(1):57. doi: 10.1056/NEJM198001033020114. No abstract available. PMID 7350401
- [Background] Goel R, Majeed F, Vogel R, Corretti MC, Weir M, Mangano C, White C, Plotnick GD, Miller M. Exercise-induced hypertension, endothelial dysfunction, and coronary artery disease in a marathon runner. Am J Cardiol. 2007 Mar 1;99(5):743-4. doi: 10.1016/j.amjcard.2006.09.127. Epub 2007 Jan 11. PMID 17317385
- [Background] Handler JB, Asay RW, Warren SE, Shea PM. Symptomatic coronary artery disease in a marathon runner. JAMA. 1982 Aug 13;248(6):717-9. No abstract available. PMID 7097925
- [Background] Hellerstein HK, Moir TW. Distance running in the 1980s: cardiovascular benefits and risks. Cardiovasc Clin. 1985;15(2):75-86. PMID 3912053
- [Background] Lehtonen A, Viikari J. Coronary-artery disease in marathon runners. N Engl J Med. 1980 Jan 3;302(1):57. No abstract available. PMID 7350402
- [Background] Maron BJ, Poliac LC, Roberts WO. Risk for sudden cardiac death associated with marathon running. J Am Coll Cardiol. 1996 Aug;28(2):428-31. doi: 10.1016/0735-1097(96)00137-4. PMID 8800121
- [Background] Mohlenkamp S, Bose D, Mahabadi AA, Heusch G, Erbel R. On the paradox of exercise: coronary atherosclerosis in an apparently healthy marathon runner. Nat Clin Pract Cardiovasc Med. 2007 Jul;4(7):396-401. doi: 10.1038/ncpcardio0926. PMID 17589430
- [Background] Mohlenkamp S, Schmermund A, Kroger K, Kerkhoff G, Brocker-Preuss M, Adams V, Hensel M, Kiefer D, Lehmann N, Moebus S, Leineweber K, Elsenbruch S, Barkhausen J, Halle M, Hambrecht R, Siegrist J, Mann K, Budde T, Jockel KH, Erbel R. Coronary atherosclerosis and cardiovascular risk in masters male marathon runners. Rationale and design of the "marathon study". Herz. 2006 Sep;31(6):575-85. doi: 10.1007/s00059-006-2879-6. PMID 17036189
- [Background] Neilan TG, Januzzi JL, Lee-Lewandrowski E, Ton-Nu TT, Yoerger DM, Jassal DS, Lewandrowski KB, Siegel AJ, Marshall JE, Douglas PS, Lawlor D, Picard MH, Wood MJ. Myocardial injury and ventricular dysfunction related to training levels among nonelite participants in the Boston marathon. Circulation. 2006 Nov 28;114(22):2325-33. doi: 10.1161/CIRCULATIONAHA.106.647461. Epub 2006 Nov 13. PMID 17101848
- [Background] Noakes TD. Heart disease in marathon runners: a review. Med Sci Sports Exerc. 1987 Jun;19(3):187-94. PMID 3298928
- [Background] Roberts WO, Maron BJ. Evidence for decreasing occurrence of sudden cardiac death associated with the marathon. J Am Coll Cardiol. 2005 Oct 4;46(7):1373-4. doi: 10.1016/j.jacc.2005.07.008. No abstract available. PMID 16198859
- [Background] Schuchert A, Puschel K, Kupper W, Schafer H, Bleifeld W. [Sudden heart death in a long distance runner during a marathon]. Z Kardiol. 1989 Apr;78(4):276-80. German. PMID 2735089
- [Background] Rowe WJ. A world record marathon runner with silent ischemia without coronary atherosclerosis. Chest. 1991 May;99(5):1306-8. doi: 10.1378/chest.99.5.1306. PMID 2019205
- [Background] Tunstall Pedoe DS. Marathon cardiac deaths : the london experience. Sports Med. 2007;37(4-5):448-50. doi: 10.2165/00007256-200737040-00046. PMID 17465632
- See also: The Minneapolis Heart Institute Foundation improves cardiovascular health through clinical research and education — http://www.mplsheart.org/
- See also: The Minneapolis Heart Institute® is recognized internationally as one of the world's leading providers of heart and vascular care — http://www.mplsheart.com